CLINICAL TRIAL: NCT02810171
Title: Dimensional Brain Behavior Predictors of CBT Outcomes in Pediatric Anxiety
Acronym: Anxiety-CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Ohio State University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Christopher Monk, Associate Chair, Department of Psychology, Professor of Psychology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00118950; R01MH107419 (NIH)
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Last update posted 2021-12-20 (Actual); Status verified 2021-07

CONDITIONS: Anxiety Disorders; Social Anxiety Disorder; Social Phobia; Generalized Anxiety Disorder; Separation Anxiety Disorder; Specific Phobia; Phobia; Agoraphobia; Panic Disorder; Panic Attack; Anxiety
Keywords: anxiety; social anxiety disorder; generalized anxiety disorder; phobias; fears; worry
MeSH Terms: conditions — Anxiety Disorders; Phobia, Social; Generalized Anxiety Disorder; Anxiety, Separation; Phobia, Specific; Phobic Disorders; Agoraphobia; Panic Disorder | interventions — Cognitive Behavioral Therapy; Relaxation Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive Behavioral Therapy (Active Comparator)
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Relaxation Therapy (Other)
  Interventions: Behavioral: Relaxation Therapy
- No Intervention: Healthy youth only (No Intervention): Healthy control participants, matched to gender and age with anxiety patients, will be enrolled. These healthy participants will be scanned with fMRI before and after ~16 weeks, but without any intervention (i.e., no therapy).

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — A therapy which teaches patients coping skills to manage anxiety and gradually yet repeatedly exposes patients to anxiety-provoking thoughts and situations until the anxiety habituates/diminishes.
  Other Names: CBT
  Arms: Cognitive Behavioral Therapy
Behavioral: Relaxation Therapy — An active control therapy with minimal effects on anxiety symptoms. If randomized to this therapy, participants will have the option to cross-over to CBT once the relaxation therapy arms has been completed.
  Arms: Relaxation Therapy

SUMMARY:
Anxiety is among the most prevalent, costly and disabling illnesses and tends emerge early in childhood. Cognitive behavioral therapy (CBT) is the first-line treatment for early life anxiety, but as many as 40% of young patients who receive CBT fail to get better. The proposed study will examine brain changes marking positive response to CBT for anxiety and how these changes may differ in children compared adolescents. By helping us to understand how CBT works, this study will pave the way for new treatments to stop anxiety early.

DETAILED DESCRIPTION:
Impairing anxiety affects 33% of the population by adolescence and can become chronic, leading to depression, substance abuse, school-drop out and even suicide. To reduce anxiety and prevent its sequelae, patients must be effectively treated early; yet, the first line intervention, cognitive behavioral therapy (CBT), has a heterogeneous response with 40-60% of treated patients continuing to experience impairment from residual symptoms. The reasons for variability in CBT outcomes remain poorly understood, but individual (including developmental) differences in brain-behavioral targets of CBT may contribute. This proposal addresses two primary questions: 1) Do individual differences in CBT-relevant brain-behavioral functions lead to variation in CBT outcomes? and 2) Does development contribute to this variation? To answer these questions, this study will measure changes in brain and behavior markers of anxiety, before and after CBT, in children and adolescents across traditional, categorical anxiety disorders (e.g., social, generalized and separation anxiety disorders). Given that CBT facilitates control over fear to enable effective regulation, the investigators hypothesize that brain-behavioral markers of fear sensitivity, cognitive regulatory capacity and cognitive regulation of fear will predict and characterize mechanisms of CBT effect. In addition, the investigators hypothesize that these markers will differentially relate to CBT effect, depending on patient age.

Children and adolescents (7.0 - 17.99 years) with clinically impairing anxiety will be randomized to receive CBT or a relaxation control therapy for 12 weeks. Before and after therapy, all participants will receive an MRI scan to see what regions of the brain become active when emotion and concentration tasks are performed and how that activation is changed after CBT.

While the study itself is of parallel design for its data-collection and measurement purpose, it is listed as a partial-crossover design in the IRB-approved protocol because subjects randomized to the relaxation therapy are given the option of receiving 12-weeks of CBT sessions after the relaxation therapy data has been collected. Some limited data will be collected in patients who are initially randomized to relaxation therapy but then opt to crossover to CBT. MRI data will also be collected in healthy youth before and after 12 weeks (but without intervening therapy) to allow the investigators to control for the simple effects of time that may cause brain changes that are not related to therapy.

ELIGIBILITY:
Inclusion Criteria for all participants (Clinically Anxious and Healthy):

* Age 7.0 - 17.99 years
* Parent or guardian able and willing to give informed consent
* Ability to tolerate small, enclosed spaces

Exclusion criteria for all participants (Clinically Anxious and Healthy)

* No metals, implants or metallic substances within or on the body (e.g., orthodontic braces)
* Vision equal to or better than 20/30 on a Snelling chart, with correction if necessary
* Not currently taking any psychotropic medication or receiving any psychotherapy (stable doses of stimulants allowable for anxiety subjects with comorbid attention deficit hyperactivity disorder) or receiving hormone therapy other than birth control
* No lifetime diagnoses of psychotic disorder, mental retardation or autism
* No history of current substance/alcohol abuse/dependence
* No evidence of suicidal intentions or behaviors in the past 6 months
* No history of serious medical or neurological illness
* If post-pubertal female, not pregnant

Additional Inclusion Criteria for Clinically Anxious Participants:

* Clinically significant anxiety as determined by structured clinical interview
* Past history of major depressive episodes are allowable
* Past history substance/alcohol abuse allowable if in remission for at least 1 year
* Obsessive-compulsive disorder symptoms are acceptable if not the primary source of interference or distress
* Anxiety must be primary concern, still bothersome, and CBT for anxiety determined to be appropriate treatment

Additional exclusion criteria for Healthy Participants:

* No history of past or current mental illness as determined by structured clinical interview

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 207 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2021-07 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
Brain function/structure as assessed by Magnetic Resonance Imaging scans | Baseline and 12-weeks
  Pre- to post-CBT changes in functional, connectivity and structural MRI measures of brain networks relevant for anxiety. Brain regions include the amygdala, anterior insula, dorsal anterior cingulate cortex (dACC) and ventrolateral prefrontal cortex (vlPFC). Functional activation and connectivity of these brain regions are assessed using simple computer tasks performed during MRI scanning. Tasks engage threat reactivity, self-regulatory control and the interaction of these processes. Structural connections between regions will be measured using a MRI technique that measures water diffusion in the brain.

SECONDARY OUTCOMES:
Pediatric Anxiety Rating Scale | weeks 0, 3, 6, 9, 12
  The Pediatric Anxiety Rating Scale (PARS) is a clinician-administered assessment to rate the severity of anxiety symptoms associated with common DSM-V anxiety disorders (social phobia, separation anxiety disorder, and generalized anxiety disorder) in children. The investigators are looking for decreases in anxiety severity ratings from pre- to post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kate D. Fitzgerald, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be shared with the National Database for Autism Research (NDAR) and the Research Domain Criteria Database (RDoCdb).

REFERENCES:
- [Derived] Diaz DE, Becker HC, Hardi FA, Beltz AM, Bilek EL, Russman Block S, Phan KL, Monk CS, Fitzgerald KD. Connectivity between the central executive and salience networks normalizes with exposure-focused CBT in pediatric anxiety. medRxiv [Preprint]. 2026 Jan 30:2026.01.28.26345061. doi: 10.64898/2026.01.28.26345061. PMID 41646716
- [Derived] Bilek EL, Iturra-Mena AM, Becker HC, Phan KL, Monk CS, Fitzgerald KD. Exposure-Focused Cognitive-Behavioral Therapy for Youth Anxiety Disorders: Superiority Over Relaxation-Based Comparator and Predictors of Response. JAACAP Open. 2025 Apr 25;3(4):1161-1176. doi: 10.1016/j.jaacop.2025.04.003. eCollection 2025 Dec. PMID 41367992
- [Derived] Diaz DE, Russman Block SR, Becker HC, Phan KL, Monk CS, Fitzgerald KD. Neural Substrates of Emotion Processing and Cognitive Control Over Emotion in Youth Anxiety: An RDoC-Informed Study Across the Clinical to Nonclinical Continuum of Severity. J Am Acad Child Adolesc Psychiatry. 2025 Apr;64(4):488-498. doi: 10.1016/j.jaac.2024.06.010. Epub 2024 Jul 24. PMID 39059719
- [Derived] Rueppel M, Mannella KA, Fitzgerald KD, Schroder HS. Post-error slowing in anxiety and obsessive-compulsive disorders. Cogn Affect Behav Neurosci. 2022 Jun;22(3):610-624. doi: 10.3758/s13415-021-00976-9. Epub 2021 Dec 29. PMID 34966981